CLINICAL TRIAL: NCT06525493
Title: Comparison of Combination of Proximal Adductor Canal Block and Infiltration Between Popliteal Artery and Capsule of Knee With Large-Volume Distal Adductor Canal Block in Facilitating Early Mobilization After Total Knee Replacement
Brief Title: Comparison of Combination of Proximal ACB and iPACK With Large-Volume Distal ACB for Early Mobilization After TKR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Pryambodho Pryambodho, dr, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 585/UN2.F1/ETIK/PPM.00.02/2023
Record Dates: First submitted 2024-07-24; First posted 2024-07-29 (Actual); Last update posted 2024-07-29 (Actual); Status verified 2024-07

CONDITIONS: Adductor Canal Block; Postoperative Pain; Regional Anesthesia
Keywords: Total Knee Replacement; Adductor Canal Block; Postoperative Pain; Regional Anesthesia; Postoperative Mobilization; TUG Test
MeSH Terms: conditions — Pain, Postoperative | interventions — Anesthesia, Conduction

STUDY DESIGN:
Who Masked: Participant
Masking Description: Single blind
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Patients receive the large-volume distal adductor canal block (ACB). In this technique, a linear transducer is placed on the medial aspect, approximately one fourth of the distal thigh to identify the Adductor Hiatus, and the injection is performed in-plane near that point using ropivacaine.
  Interventions: Procedure: Regional Anesthesia
- Group B (Experimental): This arm involves a combination of two regional anesthesia techniques: proximal adductor canal block (ACB) and iPACK. In proximal ACB, the transducer is placed in the middle of the thigh, and the injection is performed in-plane approximately 1-2 cm distal from a specific point. Meanwhile, in iPACK, the curvilinear transducer is positioned on the posteromedial aspect of the distal thigh, and the injection is performed between the popliteal artery and the femur
  Interventions: Procedure: Regional Anesthesia

INTERVENTIONS:
Procedure: Regional Anesthesia — The interventions are three different regional anesthesia techniques: Proximal Adductor Canal Block (ACB), iPACK (Interspace between the Popliteal Artery and the Capsule of the Posterior Knee), and Large-Volume Distal Adductor Canal Block (Large ACB distal). all three interventions were administered using ropivacaine 0.2%. However, there were differences in the volumes injected for each regional anesthesia technique. Proximal ACB: 15 mL of ropivacaine 0.2%. iPACK: 20 mL of ropivacaine 0.2%. Large ACB distal: 35 mL of ropivacaine 0.2%

SUMMARY:
Large-volume distal ACB is not superior to combination of proximal ACB and iPACK in facilitating early mobilization after TKR. Block performing time of distal ACB was significantly shorter compared to the combination of proximal ACB and iPACK

DETAILED DESCRIPTION:
Adductor Canal Block (ACB) and Infiltration between Popliteal Artery and Capsule of Knee (iPACK) are popular block methods for analgesia after Total Knee Replacement (TKR), covering both anterior and posterior knee. Adductor canal serves as a passageway, local anesthetic injected here will spread both to proximal and distal to posterior. Study was a single-blinded, randomized controlled trial between June 2023 and January 2024. Large-volume distal ACB is not superior to combination of proximal ACB and iPACK in facilitating early mobilization after TKR. Block performing time of distal ACB was significantly shorter compared to the combination of proximal ACB and iPACK

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 50 - 80 years who underwent total knee replacement surgery

Exclusion Criteria:

* Systemic allergy, anaphylactic reaction, and occurrence of cardiac arrest
* Intraoperative fracture
* Change to general anesthesia
* Patient who decides to withdraw from the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2024-01-01 (Actual)

PRIMARY OUTCOMES:
Timed Up and Go test on Postoperative Day 1 (POD 1) | The test is conducted specifically on the first day after the surgery, known as Postoperative Day 1 (POD 1)
  The Timed Up and Go (TUG) test is a functional mobility assessment used to evaluate a person's ability to stand up from a chair, walk a short distance, turn around, return to the chair, and sit down again. It assesses balance, gait, and functional mobility, which are crucial aspects of postoperative recovery.
Numeric Rating Scale | The NRS assessments are conducted at 6 hours, 12 hours, and 24 hours after the surgery
  The NRS is a commonly used tool to assess pain intensity. Patients are typically asked to rate their pain on a numerical scale from 0 to 10, where 0 represents no pain and 10 represents the worst imaginable pain
Total 24 hours morphine consumption | The measurement is taken over the entire 24-hour period following the surgery
  This measures the total amount of morphine consumed by patients within the first 24 hours after surgery. It reflects the effectiveness of pain management strategies and the need for opioid analgesia

CONTACTS AND LOCATIONS:
Locations (1):
- Cipto Mangunkusumo Hospital, Jakarta Pusat, DKI Jakarta, Indonesia, Jakarta Pusat, DKI Jakarta, Indonesia